CLINICAL TRIAL: NCT03095313
Title: 18-F Sodium Fluoride (18F-NaF) Positron Emission Tomography (PET) for the Assessment of Bioprosthetic Aortic Valve Durability and Outcomes
Brief Title: 18-F Sodium Fluoride (18F-NaF) PET for the Assessment of Bioprosthetic Aortic Valve Durability and Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Daniel S. Berman, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 46429
Record Dates: First submitted 2017-03-24; First posted 2017-03-29 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2022-03

CONDITIONS: Aortic Stenosis
Keywords: Transcatheter Aortic Valve Replacement (TAVR).; Surgical bioprosthetic aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 18F-NaF PET and CT scanning (Experimental): 18F-NaF PET-CT scan (at Baseline visit only) Contrast-enhanced CT Scan (at Baseline and Year 2 only) with possible beta-blocker and nitroglycerin, if medically safe.
  Interventions: Other: 18F-NaF

INTERVENTIONS:
Other: 18F-NaF — At baseline a target dose of 125 MBq 18F-NaF will be administered intravenously to all subjects who will then undergo dual cardiac and respiratory-gated PET-CT imaging of the heart and aortic valve. 125ml of iodine-based contrast agent (iohexol [Omnipaque™]) will be given for the CT. Nitroglycerin will be given to increase the size of the coronary arteries and a possible dose of metoprolol may be given to control target heart rate.
  Repeat contrast-enhanced CT of the heart and aortic valve will be conducted at Year 2 to investigate to investigate whether 18F-NaF activity predicts progression of calcification in prosthetic valves.
  Other Names: 18F Sodium Flouride; sodium flouride PET

SUMMARY:
This is a pilot study in which we will aim to demonstrate successful execution of the imaging protocol and to make observations regarding the calcification activity as measured by 18F-NaF PET/CT and any correlation to 1) valve age and valve type, and 2) subsequent degeneration of aortic valve bioprostheses based upon clinical, echocardiographic and CT parameters.

Additionally, the data will serve as preliminary data to plan a larger study to investigate study objectives.

DETAILED DESCRIPTION:
This five-year pilot study will aim to demonstrate successful execution of the imaging protocol and to make observations regarding the calcification activity as measured by 18F-NaF PET/CT and any correlation to 1) valve age and valve type, and 2) subsequent degeneration of aortic valve bioprostheses based upon clinical, echocardiographic and CT parameters. Techniques that can identify specific increases in calcification activity are therefore likely to provide important insights into predicting the longevity of TAVR valves and guidance towards subsequent interventions.

Twenty patients whom have undergone either TAVR or surgical bioprosthetic aortic valve replacement will be invited to participate in an 18F-NaF PET scan (baseline) and CT scan imaging (baseline and Year 2). Baseline, Year 1 and 2 will also include clinical assessment, labs and echocardiograms. Telephone contact at Years 3, 4, and 5 will provide follow up for major cardiovascular adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥60 years
* Patients between 1 month and 5 years following transcatheter aortic valve replacement (TAVR) or surgical bioprosthetic aortic valve replacement

Exclusion Criteria:

* Inability to provide informed consent
* Creatinine >1.5 mg/dL
* History of severe allergy to iodine contrast agents
* Active atrial fibrillation
* Paget's disease
* Metastatic malignancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-23 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Presence of calcification activity within the replacement valve by 18F-NaF PET-CT | Baseline
  Presence of calcification activity will be determined by presence of uptake of the radiotracer, 18F-NaF, on 18F-NaF PET-CT images.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Berman, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No